CLINICAL TRIAL: NCT07054203
Title: The Effects of Using Water Flosser Versus Interdental Brush on Gingival Health in Patients With Mandibular Bonded Retainer - A Randomized Controlled Trial
Brief Title: The Effects of Using Water Flosser Versus Interdental Brush on Gingival Health in Patients With Mandibular Bonded Retainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-8799-26054
Record Dates: First submitted 2025-06-25; First posted 2025-07-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Gingival Health
Keywords: fixed orthodontic treatment; gingival health; mandibular bonded retainer; water flosser; interdental brushes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Water Flosser (Experimental): This arm assigns participants to a powered Water Flosser (e.g., Waterpik Aquarius) because hydrodynamic shear forces can penetrate subgingival niches. Each participant receives standardized instruction plus a live demonstration; they then perform once-daily full-mouth irrigation for six months in addition to conventional tooth-brushing.
  Interventions: Device: Interdental Brush
- Interdental Brush (Active Comparator): Participants allocated to this arm receive Interdental Brushes matched to embrasure size. They are instructed to perform once-daily mechanical cleaning of every interproximal space for six months, again paired with twice-daily manual tooth-brushing
  Interventions: Device: Water Flosser

INTERVENTIONS:
Device: Water Flosser — Participants in this Arm used a powered oral irrigator delivering a pulsed water stream at 50-90 psi. The intervention consisted of once-daily full-mouth irrigation, added to routine tooth brushing, for a duration of six months.
  Arms: Interdental Brush
Device: Interdental Brush — Participants in this Arm used cylindrical, color-coded interdental brushes matched to individual embrasure sizes. The intervention involved once-daily cleaning of all interproximal spaces for six months, in addition to routine twice-daily tooth brushing.
  Arms: Water Flosser

SUMMARY:
This randomized controlled trial aimed to investigate and compare the effects of employing a water flosser versus an interdental brush on the gingival health of individuals with mandibular bonded retainers. The study recognized the significance of oral hygiene for individuals with such retainers, as they can pose challenges in maintaining optimal gum health due to their intricate structure. Participants were randomly allocated to either the water flosser group or the interdental brush group, and their gingival health was monitored over the course of the trial.

By evaluating key indicators of gingival health, such as plaque accumulation, bleeding, and inflammation, this study sought to shed light on the relative effectiveness of these two oral hygiene methods. The project's findings are anticipated to provide crucial insights into the most suitable and efficacious approach for individuals with mandibular bonded retainers, ultimately contributing to improved oral health outcomes and enhanced patient care. This research not only addresses a practical concern in dental care but also contributes to the broader understanding of oral hygiene strategies for patients with specialized orthodontic devices.

DETAILED DESCRIPTION:
After the removal of orthodontic appliances, retention is one of the most important aspects of orthodontic therapy Removable and fixed retainers are examples of retention appliances that have been introduced. Since their inception in 1970, bonded fixed retainers have become more popular. Fixed retainers have benefits of demanding minimal patient compliance, being unnoticeable, ensuring safe and efficient permanent retention. However; some disadvantages of fixed retainers have also been noted, including increased chair side time, technique sensitivity, possible detrimental effects on periodontal tissues, the risk for tooth displacement due to wire distortion and frequent bond failures. Fixed retainers have benefits of demanding minimal patient compliance, being unnoticeable, ensuring safe and efficient permanent retention. However; some disadvantages of fixed retainers have also been noted, including increased chair side time, technique sensitivity, possible detrimental effects on periodontal tissues, the risk for tooth displacement due to wire distortion and frequent bond failures.

Despite all the disadvantages of fixed retainers, this type of retainer has become increasingly popular and at the same time raises concerns among dentists about possible periodontal health issues. It is stated that fixed retainers are conducive for plaque retention which cause gingivitis and periodontitis. A study on fixed retainers also concluded that long-term fixed retainer wear leads to increased calculus accumulations, marginal recession, and probing depths. These effects are due to long-term tissue irritation caused by the fixed retainer and bacterial build up around it. Bonding of the retainer to each tooth may limit toothbrush access to interdental areas, decreasing the ability of floss to glide smoothly across the teeth, resulting in a decrease in overall oral hygiene maintenance of patients.

One of those cleaning devices is a water flosser, which is effective in cleaning inaccessible areas which present commonly in patients with fixed retainers and can be used to improve their gingival health. To the best of our knowledge, there has been no previous research on this subject. Therefore, the goal of this randomized controlled trial is to compare the effects of water flosser versus interdental brush in improving gingival health in patients with mandibular permanent retainers by detecting differences in debris accumulation, plaque and calculus formation, and signs of gingival inflammation such as gingival bleeding.

RATIONALE:

With the increasing usage of bonded retainers in orthodontic treatment, the concerns about their effects on periodontal health are also increasing.14 Fixed retainers' applications in orthodontics without proper interdental cleaning aids may result in inadequate oral hygiene. Therefore, it is crucial to determine effective aids that not only improve the periodontal health but also prove to be simple and efficient to use for the patients. Moreover, to the best of our knowledge, no previous study has compared the effects of water flosser and interdental brush usage on oral hygiene maintenance in patients with fixed bonded retainers. .

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing fixed orthodontic treatment requiring bonded retention
* All patients who will sign the informed consent form

Exclusion Criteria:

* • Patients with systemic diseases or multiple co-morbid such as diabetes, blood dyscrasias, etc.

  * Patients with any previous history of periodontal surgery
  * Patients with uncontrolled periodontal disease
  * Pregnant women or lactating mothers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-14 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Mean plaque scores | 6 months
  A randomized controlled trial will be carried out to compare the effects of water flosser versus interdental brush in improving gingival health in patients with mandibular permanent retainers by detecting differences in debris accumulation, plaque and calculus formation, and signs of gingival inflammation such as gingival bleeding. For this we will divide our study participants into two groups, they will be randomly allocated in Group 1: Water flosser or Group 2: Interdental brush. Both groups will undergo retention procedure as per standard protocol by bonding of retainer on lingual surfaces of lower teeth. Plaque scores will be measured thrice, once immediately after debonding followed by three months and six months after debonding using periodontal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
No data will be shared to retain patient confidentiality